CLINICAL TRIAL: NCT06039995
Title: The Efficacy of Adjuvant Oral Care in Prevention of Ventilator Associated Pneumonia: A Randomized Controlled Trial.
Brief Title: The Efficacy of Adjuvant Oral Care in Prevention of Ventilator Associated Pneumonia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Akash Samuel, Principal Investigator, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAP RCT 23
Record Dates: First submitted 2023-09-10; First posted 2023-09-15 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Pneumonia, Ventilator-Associated
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Adjuvant Oral Care) Intervention Group (Experimental): This group represents the intervention arm of the study. Patients in this arm receive a combination of interventions, including Chlorhexidine mouthwash, toothbrushing, and the application of moisturizing gel on the interior and exterior surfaces of the oral cavity. This group is the focus of the study's investigation to determine the effectiveness of adjuvant oral care in reducing the incidence of Ventilator-Associated Pneumonia (VAP) and improving patient outcomes.
  Interventions: Procedure: Comprehensive Oral Care; Device: Mechanical Tooth Brushing using 0.2% Chlorhexidine; Device: Moisturizing Gel
- (Traditional Oral Care) Control Group (Active Comparator): This group represents the control arm of the study. Patients in this arm receive traditional oral care, which involves the use of 0.2% Chlorhexidine mouthwash only.
  Interventions: Procedure: Traditional Oral Care; Device: Oral care using Cotton swab dipped in 0.2% Chlorhexidine

INTERVENTIONS:
Procedure: Comprehensive Oral Care — The intervention mentioned in this study involves a combination of oral care strategies for patients in the intervention group. These strategies include:
  Chlorhexidine Mouthwash: Patients in the intervention group will receive Chlorhexidine mouthwash. Chlorhexidine is known for its effectiveness in maintaining oral hygiene.
  Toothbrushing: In addition to Chlorhexidine mouthwash, patients in the intervention group will undergo toothbrushing. This involves cleaning the teeth and surrounding oral tissues to ensure thorough oral hygiene.
  Moisturizing Gel Application: The intervention group will also receive the application of moisturizing gel on the interior and exterior surfaces of the oral cavity. This helps in maintaining the moisture content of the oral tissues.
  These interventions aim to enhance oral care beyond traditional methods, potentially reducing the risk of Ventilator-Associated Pneumonia (VAP) and improving overall patient outcomes in the intensive care unit (ICU).
  Other Names: Adjuvant oral care as a component of traditional oral care
  Arms: (Adjuvant Oral Care) Intervention Group
Procedure: Traditional Oral Care — In the control arm, patients receive the intervention known as "Traditional Oral Care." This involves the use cotton swab dipped in 0.2% Chlorhexidine mouthwash for oral hygiene.
  Arms: (Traditional Oral Care) Control Group
Device: Mechanical Tooth Brushing using 0.2% Chlorhexidine — Toothbrushing: In addition to Chlorhexidine mouthwash, patients in the intervention group will undergo toothbrushing. This involves cleaning the teeth and surrounding oral tissues to ensure thorough oral hygiene.
  Arms: (Adjuvant Oral Care) Intervention Group
Device: Moisturizing Gel — Moisturizing Gel Application: The intervention group will also receive the application of moisturizing gel on the interior and exterior surfaces of the oral cavity. This helps in maintaining the moisture content of the oral tissues.
  Other Names: Veramin
  Arms: (Adjuvant Oral Care) Intervention Group
Device: Oral care using Cotton swab dipped in 0.2% Chlorhexidine — This involves the use cotton swab dipped in 0.2% Chlorhexidine mouthwash for oral hygiene
  Arms: (Traditional Oral Care) Control Group

SUMMARY:
A Randomized Controlled Trial (RCT) at Services Hospital, Lahore, aims to reduce Ventilator-Associated Pneumonia (VAP) incidence and mortality rates while shortening ICU stays in mechanically ventilated patients by adding adjuvant oral care to traditional practices.

Study Objectives:

Focus: ICU patients on mechanical ventilation. Question: Does adjuvant oral care reduce VAP rates and ICU stays?

Methodology:

Sample: Minimum 100 eligible subjects via convenient sampling. Randomization: Computer software for unbiased group allocation. Interventions: Intervention group gets Chlorhexidine mouthwash, toothbrushing, and oral gel; control group gets 0.2% Chlorhexidine mouthwash.

Measures: Evaluate VAP using Modified Clinical Pulmonary Infection Score (MCPIS) and compare demographic data.

Statistical Analysis: SPSS v22 to analyze data.

Expected Impact:

Potential to reduce VAP and improve ICU patient outcomes. Cost-effective treatment with adjuvant oral care. Shorter ICU stays, relieving VAP burden. Enhanced patient care, reduced mortality, and resource strain. Aligns with reducing VAP incidence and improving ICU patient care.

DETAILED DESCRIPTION:
The study in question is a Randomized Controlled Trial (RCT) conducted at Services Hospital, Lahore, over a three-month duration. It aims to assess the effects of including adjuvant oral care as part of traditional oral care in reducing the incidence and mortality rates of Ventilator-Associated Pneumonia (VAP) while also shortening the length of ICU stays among patients on mechanical ventilation. This research holds the potential to bring significant improvements to patient care and reduce the burden of VAP in critical care settings.

Study Objectives:

Population Focus: The study focuses on patients admitted to the intensive care unit (ICU) who are receiving mechanical ventilation.

Research Question: The central question this study seeks to answer is: Does the inclusion of adjuvant oral care alongside traditional oral care reduce the incidence and mortality rates of VAP and shorten the length of ICU stay among patients on mechanical ventilation?

Methodology:

Sample Selection: The study aims to include a minimum of 100 subjects who meet the inclusion criteria. These subjects will be selected through convenient sampling.

Randomization: To ensure unbiased allocation, subjects will be randomly assigned to either the control group or the intervention group using computer software.

Interventions: The intervention group will receive a combination of interventions, including Chlorhexidine mouthwash, toothbrushing, and the application of moisturizing gel on the interior and exterior surfaces of the oral cavity. In contrast, the control group will receive traditional oral care involving the use of 0.2% Chlorhexidine mouthwash only.

Outcome Measures: The study will evaluate the incidence of VAP by employing the Modified Clinical Pulmonary Infection Score (MCPIS). Additionally, demographic characteristics such as age, gender, smoking history, duration of ICU stay, and mortality rates will be compared between the two groups.

Statistical Analysis: Data analysis will be conducted using SPSS version 22, employing appropriate statistical methods and tests to draw meaningful conclusions.

Expected Impact:

The findings of this study hold significant potential to reduce VAP rates and improve patient outcomes in ICU settings. The incorporation of toothbrushing and moisturizing gel alongside Chlorhexidine mouthwash may enhance the cost-effectiveness of treatment and benefit healthcare professionals. This approach could potentially lead to shorter ICU stays, ultimately reducing the burden of VAP in critical care settings.

Furthermore, the implementation of comprehensive oral care practices beyond traditional methods has the potential to improve patient care, decrease mortality rates, and alleviate the strain on healthcare resources by potentially reducing the duration of ICU stays. In sum, this research contributes to the broader goal of reducing the incidence of VAP and enhancing overall patient care in intensive care units.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients on intensive mechanical ventilation aged 18-65 years of either sex with oral ETT in situ.
* MCPIS score between 0 to 5 on first day of admission at ICU

Exclusion Criteria:

* More than 48 hours of mechanical ventilation before ICU admission.
* Previous history of respiratory illness.
* Immunocompromised.
* Ongoing sepsis.
* Pregnancy.
* Presence of dentures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akash Samuel, MS Nursing, Principal Investigator — University of Health Sciences Lahore
Locations (2):
- Pakistan (2):
  - University of Health Sciences, Lahore, Punjab Province
  - Services Hospital, Lahore

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- (Adjuvant Oral Care) Intervention Group: The intervention arm of the study focuses on evaluating the effectiveness of comprehensive oral care in reducing Ventilator-Associated Pneumonia (VAP) and improving patient outcomes. Patients in this group receive a combination of interventions, including Chlorhexidine mouthwash, toothbrushing, and moisturizing gel application.
  The oral care strategies include:
  Chlorhexidine Mouthwash: Known for its role in maintaining oral hygiene, this antiseptic rinse helps reduce bacterial load in the oral cavity.
  Toothbrushing: Mechanical toothbrushing using 0.2% Chlorhexidine ensures thorough cleaning of teeth and surrounding tissues, enhancing oral hygiene.
  Moisturizing Gel Application: Applied to both interior and exterior oral surfaces, this gel helps maintain moisture levels and prevent tissue dryness.
  These interventions go beyond standard oral care, aiming to minimize the risk of VAP and improve patient health in the ICU.
Period: Overall Study
Arm/Group | (Adjuvant Oral Care) Intervention Group | (Traditional Oral Care) Control Group
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | (Adjuvant Oral Care) Intervention Group | (Traditional Oral Care) Control Group | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.71 (10.54) | 48.83 (11.6) | 48.77 (11.025)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 25 | 26 | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 50 | 50 | 100
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Pakistan | 50 | 50 | 100
Number of Participants with Ventilator Associated Pneumonia [Count of Participants; unit: Participants] | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Ventilator-Associated Pneumonia (VAP)
Description: This outcome measures the number of participants who developed ventilator-associated pneumonia (VAP) within the early period following initiation of mechanical ventilation. VAP was assessed using clinical and diagnostic criteria on the fifth day after implementation of the assigned oral care intervention. This outcome was used to evaluate the effectiveness of adjuvant oral care compared with traditional oral care in preventing early-onset VAP.
Time Frame: Five days after initiation of the assigned oral care intervention.
Measure: Count of Participants; unit: Participants
Groups:
- (Adjuvant Oral Care) Intervention Group: This group constitutes the intervention arm of the study. Patients assigned to this arm receive comprehensive oral care consisting of chlorhexidine mouthwash, mechanical toothbrushing, and application of moisturizing gel to both the interior and exterior surfaces of the oral cavity. The purpose of this intervention is to evaluate the effectiveness of enhanced oral care as an adjunct strategy in reducing the incidence of ventilator-associated pneumonia (VAP) and improving patient outcomes in the intensive care unit (ICU).
  Components of the Intervention
  Chlorhexidine Mouthwash (0.2%) Patients receive 0.2% chlorhexidine mouthwash, an established antimicrobial agent used to reduce oral microbial load and maintain oral hygiene.
  Mechanical Toothbrushing Toothbrushing is performed to mechanically remove dental plaque and debris from the teeth and surrounding oral tissues, ensuring thorough oral hygiene beyond chemical disinfection alone.
  Moisturizing Gel Application A moisturizing gel is applied to the interior and exterior surfaces of the oral cavity to prevent oral dryness and maintain mucosal integrity.
  Together, these interventions provide a comprehensive oral care regimen designed to enhance standard care practices, reduce bacterial colonization, and potentially lower the risk of VAP while improving overall patient comfort and clinical outcomes.
Arm/Group | (Adjuvant Oral Care) Intervention Group | (Traditional Oral Care) Control Group
Number analyzed (Participants) | 50 | 50
Participants | 16 | 27

2. Secondary Outcome: Duration of ICU Stay
Description: The duration of ICU stay will be recorded for each patient. This data will help evaluate whether the intervention affects the length of ICU stay and potentially reduces healthcare resource utilization
Time Frame: These demographic characteristics and clinical parameters will be assessed throughout the three-month duration of the study at Services Hospital, Lahore.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | (Adjuvant Oral Care) Intervention Group | (Traditional Oral Care) Control Group
Number analyzed (Participants) | 50 | 50
Days | 12.28 (7.15) | 11.19 (6.97)

3. Secondary Outcome: Mortality Rates
Description: Mortality rates in both the control and intervention groups will be compared to assess if the adjuvant oral care intervention has an impact on patient survival during their ICU stay.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | (Adjuvant Oral Care) Intervention Group | (Traditional Oral Care) Control Group
Number analyzed (Participants) | 50 | 50
Participants | 22 | 33

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- (Adjuvant Oral Care) Intervention Group: This group represents the intervention arm of the study. Patients in this group receive comprehensive oral care consisting of 0.2% chlorhexidine mouthwash, mechanical toothbrushing, and application of a moisturizing gel to the interior and exterior surfaces of the oral cavity.
  The intervention is designed to enhance standard oral hygiene practices by reducing oral microbial load, removing dental plaque, and maintaining oral mucosal moisture. Chlorhexidine mouthwash provides antimicrobial action, while mechanical toothbrushing ensures effective removal of debris and plaque from teeth and surrounding tissues. The application of moisturizing gel helps prevent oral dryness and preserves mucosal integrity.
  This combined oral care regimen is implemented to evaluate its effectiveness as an adjuvant measure in reducing the incidence of ventilator-associated pneumonia (VAP) and improving overall patient outcomes in the intensive care unit (ICU).
Arm/Group | (Adjuvant Oral Care) Intervention Group | (Traditional Oral Care) Control Group
All-Cause Mortality (participants affected / at risk) | 22/50 | 33/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2025-12-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT06039995/Prot_000.pdf
  • Statistical Analysis Plan (2025-12-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT06039995/SAP_001.pdf